CLINICAL TRIAL: NCT00746655
Title: A Study of Stereotactic Body Radiation Therapy (SBRT) in Combination With Cisplatin Transcatheter Arterial Chemoembolization (TACE) for Primary Hepatocellular Carcinoma (HCC)
Brief Title: SBRT + TACE for Primary Hepatocellular Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dwight Heron, Vice Chairman of Clinical Affairs, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-042
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT / TACE (Other)
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Transcatheter Arterial Chemoembolization (TACE)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — The first four patients will receive 50 Gy in 5 fractions (10 Gy /fx) over a 2 week period. The next four patients will be treated to a total dose of 60 Gy in 5 fractions (15 Gy/fx) over two weeks. The final four patients will receive 75 Gy in 5 fractions (15 Gy/fx) delivered over a 2-week period,
  Other Names: CyberKnife; Trilogy
Procedure: Transcatheter Arterial Chemoembolization (TACE) — . Intra-arterial cisplatin treatment will be given at a dose of 125 mg/m2. After delivery of the drug(s) to the tumor, embolization will be accomplished with Embospheres (Biosphere Medical, Inc.,Rockland, MA, USA) until moderate to marked stasis of antegrade flow is seen in the artery.
  Other Names: Cisplatin

SUMMARY:
The purpose of this study is to determine the feasibility and toxicity of combining SBRT and TACE for unresectable HCC and to evaluate the Health Related Quality of Life (HRQL) associated with combined therapy.

DETAILED DESCRIPTION:
Patients who are poor surgical candidates could potentially benefit from non-surgical alternatives such as stereotactic body radiation therapy (SBRT). SBRT is an ideal approach to minimize radiation exposure to the normal liver while maximizing the dose to the tumor. Transarterial chemoembolization (TACE) is the combined use of intra-arterial chemotherapy and particulate arterial embolization. This technique is typically used to make unresectable liver lesions amenable to resection, for palliation in cases of extra-hepatic spread or recurrence, or for symptomatic relief. The combination of intraarterial chemotherapy with vessel embolization makes logical sense since primary and secondary liver tumors derive up to 95% of their blood supply from the hepatic artery, while the normal liver gains the majority of its blood supply from the portal system. Thus, using transarterial chemoembolization it is possible to achieve high intratumor drug concentrations followed by local ischemia, allowing uninvolved liver to be spared. This study is to determine that these standard of care therapies combined to improve the quality of life for the patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. A life expectancy of at least 12 weeks with a Karnofsky performance status of at least 70 (Appendix III)
3. HCC confirmed by biopsy OR diagnosed by clinical and radiologic criteria. All of the following criteria must be met or a biopsy is required: • Known cirrhosis or chronic HBV or HCV infection, • Hypervascular liver masses >2 cm, and either serum AFP > 400 ng/ml, or • AFP >three times normal and doubling in value in the antecedent 3 months.
4. The target lesion(s) can be accurately measured in at least one dimension according to RECIST and must have a combined maximum tumor volume of ≤ 180 cm3.
5. No prior radiotherapy to the liver.
6. Previous systemic chemotherapy or non-radiation local therapy (such as surgery, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation) is allowed. The lesion must however have shown criteria of progression based on RECIST. Local therapy must be completed at least 4 weeks prior to the baseline scan.
7. Cirrhotic status of Child-Pugh class A or B (Appendix I)
8. Patient's lesions are deemed unresectable.
9. Patient's tumor burden or medical comorbidities disqualify them for transplant OR the patient qualifies for transplant but refuses the operation OR patients planned for TACE as a bridge to transplant operation.
10. Platelet count ≥ 60 x 109/L, Hemoglobin ≥ 8.5 g/dL, WBC ≥ 2000/μL International normalized ratio (INR) ≤ 1.5 or a PT/PTT within normal limits. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.
11. Other baseline labs must meet the following criteria: total bilirubin <3mg/dl, albumin>2.5mg/dl, and liver enzymes less than three times the upper limit of normal. Creatinine must also be <1.8mg/dl or a creatinine clearance >50ml/min.
12. Must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the nature of the therapy, alternatives, potential benefits, side-effects, risks and discomforts.

Exclusion Criteria:

1. Renal failure requiring hemo- or peritoneal dialysis
2. Uncontrolled inter-current illness (except Hepatitis) including, but not limited to ongoing or active infection (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0), congestive heart failure (> New York Heart Association (NYHA) class 2), active coronary artery disease (CAD), cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin), uncontrolled hypertension and any condition which could jeopardize the safety of the patient and his/her compliance in the study . Myocardial infarction more than 6 months prior to study entry is permitted.
3. A history of variceal bleeding where the varices have not been eradicated or decompressed by shunt placement.
4. History of an active connective tissue disorder.
5. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
6. Pregnant or breast-feeding patients are excluded from this study because abdominal radiation therapy has potential for teratogenic and/or abortifacient effects.
7. Total portal vein occlusion.
8. Extensive liver tumor burden, defined as more than 75% of the liver.
9. Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.
10. Patients with uncontrolled distant disease will be excluded from this protocol. Those with controlled systemic disease will still be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and toxicity of combining SBRT and TACE for HCC. | Until disease progression
To evaluate the Health Related Quality of Life (HRQL) associated with combined therapy. | Until disease progression

SECONDARY OUTCOMES:
To determine local response of combination therapy with PET/CT and CT only. | Every 8 weeks
To evaluate the progression free interval associated with this local regional therapy. | Until disease progression
To determine if SBRT and TACE will be able to bridge patients to transplant that were initially ineligible. | Until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Dwight E Heron, MD, Study Chair — University of Pittsburgh Medical Center
Locations (4):
- United States (4):
  - UPMC Presbyterian/Montifore, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - UPMC Shadyside Radiation Oncology, Pittsburgh, Pennsylvania